CLINICAL TRIAL: NCT05085002
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of Lerociclib in Participants With Advanced Breast Cancer
Brief Title: A Study of Lerociclib in Participants With Advanced Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is being closed based on corporate changes at EQRx and is not related to any efficacy or safety issues with lerociclib.
Sponsor: EQRx, Inc. (Industry)
Responsible Party: Sponsor
Organization: EQRx International, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EQ132-201
Record Dates: First submitted 2021-09-07; First posted 2021-10-20 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-12

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Letrozole; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lerociclib + letrozole or fulvestrant (Other)
  Interventions: Drug: Lerociclib + Letrozole or Fulvestrant

INTERVENTIONS:
Drug: Lerociclib + Letrozole or Fulvestrant — All participants (1L and 2L populations) will receive an AI (letrozole) or fulvestrant plus lerociclib 150 mg BID.

SUMMARY:
This is a multicenter, single-arm, open-label study to evaluate the safety and efficacy of lerociclib in combination with standard endocrine therapy in female or male participants with HR+/HER2- MBC. The study population will consist of either newly diagnosed, treatment naïve participants with HR+/HER2- MBC (1L population) and participants with HR+/HER2- MBC who have already progressed on first line endocrine therapy such as tamoxifen, anastrozole, or letrozole (2L population). All premenopausal or perimenopausal female participants, and all male participants, must be receiving goserelin for at least 28 days prior to entering the study and will remain on goserelin throughout the study, in accordance with the prescribing information and according to the study site's standard practice.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 or the legal age of consent in the jurisdiction in which the study is taking place, at the time of signing the informed consent.
2. Histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer by local laboratory and has HER2-negative breast cancer.
3. Advanced (locoregionally recurrent not amenable to curative therapy, eg, surgery and/or radiotherapy, or metastatic) breast cancer
4. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1.
5. Adequate bone marrow and organ function
6. Female that is not pregnant and agrees to contraceptive use that is consistent with local regulations regarding the methods of contraception to be used during the study
7. Males agree to use a highly effective method of contraception and will refrain from donating sperm from the first dose of any study intervention
8. Participant is capable of giving signed informed consent

Exclusion Criteria:

1. Symptomatic visceral disease or any disease burden that makes the participant ineligible for endocrine therapy per the Investigator's best judgment.
2. Peritoneal carcinomatosis.
3. Inflammatory breast cancer at screening.
4. Participant with central nervous system (CNS) involvement unless they are at least 4 weeks from prior therapy completion to starting the study treatment and have stable CNS tumor at the time of screening and not receiving steroids and/or enzyme inducing anti-epileptic medications for brain metastases.
5. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality
6. Has a history of prolonged QT syndrome or Torsades de Pointes
7. Has received prior treatment with chemotherapy (except for neoadjuvant/ adjuvant chemotherapy) or any CDK4/6 inhibitor.
8. Has received prior treatment with fulvestrant.
9. Use of systemic estrogens
10. Participant is currently receiving any of the following substances and cannot be discontinued 14 days prior to start the treatment:

    * Known strong or moderate CYP3A inducers or strong inhibition of CYP3A
    * Substances that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5.
11. Echocardiogram done within the past 12 months with ejection fraction of ≤ 45% or documented history of congestive heart failure with reduced ejection fraction.
12. Evidence of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection or oral temperature > 38°C at screening
13. Interstitial pneumonia or severe impairment of lung function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs and SAEs | Up to 4.5 years
  The number and percentage of participants experiencing any TEAE and serious TEAE will be tabulated by line of therapy.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (6):
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Oregon Oncology Specialists, Salem, Oregon
  - Cancer Care Associates of York, Inc., York, Pennsylvania
  - Tranquil Clinical Research, Webster, Texas
  - Northwest Medical Specialties PLLC, Tacoma, Washington
- Belgium (5):
  - UZA, Edegem
  - Ziekenhuizen K.U.Leuven, Campus gasthuisberg, Leuven
  - CHA Libramont, Libramont
  - Clinique Saint-Pierre asbl, Ottignies
  - vzw Verenigde Ziekenhuizen van Waas en Durme - VITAZ, Sint-Niklaas
- Georgia (5):
  - LTD "Brothers", Batumi
  - ARENSIA Exploratory Medicine LLC, Tbilisi
  - Ltd Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - LTD "Health House", Tbilisi
  - Ltd "Multiprofile Clinic Consilium Medulla ", Tbilisi
- Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori", Meldola, Italy
- Mexico (3):
  - PanAmerican Clinical Research Guadalajara, Guadalajara, Jalisco
  - PanAmerican Clinical Research Cuernavaca, Cuernavaca
  - PanAmerican Clinical Research, Queretaro, Querétaro
- IMSP Institutul Oncologic, Arsenia Exploratory Medicine, Chisinau, Moldova